CLINICAL TRIAL: NCT01652495
Title: Evaluation of Efficacy and Hypothalamus-pituitary-adrenal Axis Suppression Due to a Single Intrabursal Injection of Corticosteroids in Patients With Shoulder Calcific Tendinopathy
Brief Title: Evaluation of Efficacy and Hypothalamus-pituitary-adrenal Axis Suppression Due to Corticosteroids Intrabursal Injection
Acronym: TPESP2011-12
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Azienda Ospedaliera San Giovanni Battista (Other)
Responsible Party: Principal Investigator, milva.battaglia, Clinician, Principal Investigator, Department of Radiology, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-000866-40
Record Dates: First submitted 2012-07-21; First posted 2012-07-30 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Tendinopathy; Adrenal Insufficiency
Keywords: rotatory cuff calcific tendonitis; corticosteroids; US guided percutaneous treatment; methylprednisolone; triamcinolone; hypothalamus pituitary adrenal axis
MeSH Terms: conditions — Tendinopathy; Adrenal Insufficiency | interventions — Methylprednisolone Acetate; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- methylprednisolone acetate group (Active Comparator): Single intrabursal injection of methylprednisolone acetate
  Interventions: Drug: methylprednisolone acetate
- Triamcinolone acetonide group (Active Comparator): Single intrabursal injection of Triamcinolone acetonide
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: methylprednisolone acetate — Single intrabursal ultrasound guided injection of 40 mg (1 ml) of methylprednisolone acetate
  Other Names: Depo-medrol
  Arms: methylprednisolone acetate group
Drug: Triamcinolone Acetonide — Single intrabursal ultrasound guided injection of 40 mg (1 ml) of triamcinolone acetonide
  Other Names: Triamvirgi
  Arms: Triamcinolone acetonide group

SUMMARY:
The purpose of this study is to compare the efficacy and effects on the hypothalamus-pituitary-adrenal axis of a single intrabursal injection of two different types of corticosteroids (methylprednisolone and triamcinolone) in patients with calcific shoulder tendinopathy.

DETAILED DESCRIPTION:
Rotator cuff calcific tendonitis is a common disease, mainly affecting women aged 30 to 50 years old. It is associated to severe pain and impotence. US-guided percutaneous treatment is considered the gold standard treatment with the aim to destroy and wash out shoulder's calcification, responsible for inflammation, pain and functional limitation. Corticosteroids are injected in the subacromial-subdeltoid bursa at the end of the procedure to facilitate the prompt pain relief and functional recovery. Although corticosteroids represent the most powerful drugs to reduce inflammation and pain, their use is associated to important side effects, mainly the suppression of the hypothalamus-pituitary-axis (HPA). At the same time, no standardized protocols exist regarding the best type and dose of corticosteroid to be injected in association to the above mentioned treatment, nor data evaluating the exact duration of HPA suppression following a single intrabursal injection of corticosteroids.

40 patients affected by rotator cuff calcific tendonitis will be enrolled in the study and randomly assigned to two groups: one group (20 patients) will be treated with a single intrabursal injection of 40 mg of methylprednisolone; the other group (20 patients) will be treated with a single intrabursal injection of 40 mg of triamcinolone.

All patients will be tested at time 0 (morning before treatment) and at 1, 7, 15, 30 and 45 days after the injection, using clinical, laboratory and US parameters in order to compare the efficacy and safety of the two drugs.

ELIGIBILITY:
Inclusion Criteria:

* painful rotator cuff calcific tendonitis demonstrated by ultrasounds

Exclusion Criteria:

* pregnancy
* use of corticosteroids in the previous 2 months
* systemic chronic inflammatory or allergic diseases
* allergy to methylprednisolone or triamcinolone
* diabetes
* glaucoma
* coagulopathies or current treatment with antiaggregants or anticoagulants
* septic arthritis or infections
* calcific enthesopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Milva Battaglia, MD, Principal Investigator — Istituti Ortopedici Rizzoli
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy

REFERENCES:
- [Background] Serafini G, Sconfienza LM, Lacelli F, Silvestri E, Aliprandi A, Sardanelli F. Rotator cuff calcific tendonitis: short-term and 10-year outcomes after two-needle us-guided percutaneous treatment--nonrandomized controlled trial. Radiology. 2009 Jul;252(1):157-64. doi: 10.1148/radiol.2521081816. PMID 19561254
- [Background] Uhthoff HK, Loehr JW. Calcific Tendinopathy of the Rotator Cuff: Pathogenesis, Diagnosis, and Management. J Am Acad Orthop Surg. 1997 Jul;5(4):183-191. doi: 10.5435/00124635-199707000-00001. PMID 10797220
- [Background] Krasner AS. Glucocorticoid-induced adrenal insufficiency. JAMA. 1999 Aug 18;282(7):671-6. doi: 10.1001/jama.282.7.671. No abstract available. PMID 10517721
- [Background] Spiegel RJ, Vigersky RA, Oliff AI, Echelberger CK, Bruton J, Poplack DG. Adrenal suppression after short-term corticosteroid therapy. Lancet. 1979 Mar 24;1(8117):630-3. doi: 10.1016/s0140-6736(79)91077-8. PMID 85870
- [Background] Mader R, Lavi I, Luboshitzky R. Evaluation of the pituitary-adrenal axis function following single intraarticular injection of methylprednisolone. Arthritis Rheum. 2005 Mar;52(3):924-8. doi: 10.1002/art.20884. PMID 15751089
- [Background] Duclos M, Guinot M, Colsy M, Merle F, Baudot C, Corcuff JB, Lebouc Y. High risk of adrenal insufficiency after a single articular steroid injection in athletes. Med Sci Sports Exerc. 2007 Jul;39(7):1036-43. doi: 10.1249/mss.0b013e31805468d6. PMID 17596769

RESULTS

PARTICIPANT FLOW:
Groups:
- Methylprednisolone Acetate Group: Single intrabursal injection of methylprednisolone acetate
  methylprednisolone acetate: Single intrabursal ultrasound guided injection
- Triamcinolone Acetonide Group: Single intrabursal injection of Triamcinolone acetonide
  Triamcinolone Acetonide: Single intrabursal ultrasound guided injection
Period: Overall Study
Arm/Group | Methylprednisolone Acetate Group | Triamcinolone Acetonide Group
Started | 22 | 22
Completed | 20 | 20
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Methylprednisolone Acetate: Single intrabursal injection of 40 mg (1 ml) of methylprednisolone acetate
- Triamcinolone Acetonide: Single intrabursal injection of 40 mg (1 ml) of trimacinolone acetonide
- Total: Total of all reporting groups
Arm/Group | Methylprednisolone Acetate | Triamcinolone Acetonide | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.05 (6.67) | 46.35 (7.27) | 48.70 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 8 | 22
  Male | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Functional Improvement Measured According to Percentage Change in Constant Score
Description: Patients will be evaluated clinically by Constant Score
  Constant score: range 0 (total shoulder impairment) to 100 (non impaired shoulder). The score is obtained from two subjective (pain and relation between pain and daily-life activities) - and two objective physician-assessed (strength and range of motion) measurements
  Reference: Constant CR and Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4.
Time Frame: 180 days after treatment
Measure: Mean (95% Confidence Interval); unit: percentage of improvement Constant score
Arm/Group | Methylprednisolone Acetate Group | Triamcinolone Acetonide Group
Number analyzed (Participants) | 20 | 20
percentage of improvement Constant score | 99 [97 to 100] | 95 [93 to 97]

2. Secondary Outcome: Percentage of Patients With Suppression of Hypothalamus-pituitary-adrenal Axis
Description: Evaluation of blood cortisol and ACTH, free urinary cortisol, urinary levels of methylprednisolone or triamcinolone (depending on the administered drug) by RIA immunoassay and tandem mass assays
  Persistent suppression of the HPA axis at the end of the follow up is based on the evidence of ACTH, plasmatic and urinary cortisol levels under reference values
Time Frame: 45 days after treatment
Measure: Number; unit: % of patients with HPA suppression
Arm/Group | Methylprednisolone Acetate Group | Triamcinolone Acetonide Group
Number analyzed (Participants) | 20 | 20
% of patients with HPA suppression | 0 | 15

3. Secondary Outcome: Reduction of Pain Severity Expressed as Percentage Change in VAS Score
Description: VAS score
  VAS score is a 10 -cm graduated scale with scores ranging from 0 (no pain) to 10 (unbearable pain) self- reported by patients
  Reference: Langley GB and Sheppeard H. The visual analogue scale: its use in pain measurement. Rheumatol Int 1985;5(4):145-148.
Time Frame: 180 days after treatment
Measure: Mean (95% Confidence Interval); unit: percentage of pain reduction
Arm/Group | Methylprednisolone Acetate Group | Triamcinolone Acetonide Group
Number analyzed (Participants) | 20 | 20
percentage of pain reduction | 82 [73 to 91] | 96 [87 to 100]

ADVERSE EVENTS:
Arm/Group | Methylprednisolone Acetate Group | Triamcinolone Acetonide Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No